CLINICAL TRIAL: NCT03286881
Title: Brief Evidence-based Psychological Treatments for Emotional Disorders. A Randomized Clinical Trial in Primary and Secondary Care.
Brief Title: Brief Evidence-based Psychological Treatments for Emotional Disorders
Acronym: PsycBrief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Jorge Corpas López, Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSI2014-56368-R
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Anxiety Disorders; Depression; Somatoform Disorders; Common Mental Disorders
Keywords: Common Mental Disorders; Brief Psychological Treatments; Primary Care; Randomized Clinical Trial
MeSH Terms: conditions — Anxiety Disorders; Depression; Somatoform Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental)
  Interventions: Other: Brief individual psychotherapy
- Group 2 (Experimental)
  Interventions: Other: Brief group psychotherapy
- Group 3 (Experimental)
  Interventions: Other: Combined intervention
- Group 4 (Experimental)
  Interventions: Other: Minimum psychological intervention
- Group 5 (Active Comparator)
  Interventions: Other: Usual treatment

INTERVENTIONS:
Other: Brief individual psychotherapy — Individual brief psychological intervention by adaptation of the Guide NICE "Common Mental Health Disorders" (ISBN 978-1-84936-585-7) and the unified protocol for the trasndiagnostic treatment of the emotional disorders of Barlow (Boisseau, Farchione, Fairholme, Ellard, y Barlow, 2010). This intervention is provided by clinical psychologist in secondary care.
  Arms: Group 1
Other: Brief group psychotherapy — Group brief psychological intervention by adaptation of the Guide NICE "Common Mental Health Disorders" (ISBN 978-1-84936-585-7) and the unified protocol for the trasndiagnostic treatment of the emotional disorders of Barlow (Boisseau, Farchione, Fairholme, Ellard, y Barlow, 2010). This intervention is provided by clinical psychologist in primary care.
  Arms: Group 2
Other: Combined intervention — Traditional psychotherapy and medication provided by a clinical psychologist and a psychiatrist in secondary care.
  Arms: Group 3
Other: Minimum psychological intervention — Psychoeducation and bibliotherapy provided by a trained general practitioner in primary care.
  Arms: Group 4
Other: Usual treatment — Medication provided by a general practitioner.
  Arms: Group 5

SUMMARY:
The present work aims to develop a randomized clinical trial with a sample of 165 patients diagnosed with an emotional disorder. All participants are tested by several self-reports related to common mental disorders in a repeated measures design, pre and post treatment as well as a six month follow up. We think this study will demonstrate that brief psychological treatments should be prioritized over pharmacological treatment for such pathologies in the Primary or Secondary Care context to improve the patient´s quality of life while simultaneously reducing costs.

DETAILED DESCRIPTION:
Nowadays, the heavy demands placed on health systems exceed the resources in many developed countries. So-called "common mental disorders" and their mostly pharmacological treatment are, in no small part, responsible for this situation. The cost that these disorders generate to the public health service is very high and they are usually associated with other issues like hyperfrequentation and side effects. However, research indicates that psychological treatment should be the first step when caring for these types of problems. We expect that the results show that extensive psychological therapy and combined treatment were the most effective. Nevertheless, brief psychological treatment is expected to be the most efficient in cost-benefit terms.

ELIGIBILITY:
Inclusion Criteria:

* Emotional disorders

Exclusion Criteria:

* Severe mental disorder
* Drug abuse
* Severe depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Generalised Anxiety Disorder Assessment (GAD-7) | 12 weeks
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for GAD.
The State-Trait Anxiety Inventory (STAI) | 12 weeks
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress AnxietyForm Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level. Internal consistency coefficients for the scale have ranged from .86 to .95; test-retest reliability coefficients have ranged from .65 to .75 over a 2-month interval (Spielberger et al., 1983).
The Patient Health Questionnaire (PHQ-9) | 12 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Beck Depression Inventory-Second Edition (BDI-II) | 12 weeks
  The BDI-II is a widely used 21-item self-report inventory measuring the severity of depression in adolescents and adults. The BDI-II was revised in 1996 to be more consistent with DSM-IV criteria for depression. For example, individuals are asked to respond to each question based on a two-week time period rather than the one-week timeframe on the BDI. The BDI-II is widely used as an indicator of the severity of depression, but not as a diagnostic tool, and numerous studies provide evidence for its reliability and validity across different populations and cultural groups.
The Patient Health Questionnaire (PHQ-15) | 12 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-15 is the somatization module, which scores each DSM-IV criteria as "0" (not bothered at all) to "2" (bothered a lot).
The Patient Health Questionnaire (PHQ-PD) | 12 weeks
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.The PHQ-PD is the panic disorder module, which scores each DSM-IV criteria as "yes" or "no".
Brief Symptom Inventory 18 (BSI-18) | 12 weeks
  The BSI-18 contains the three six-item scales somatization, depression, and anxiety as well as the Global Severity Index (GSI), including all 18 items. The BSI-18 is the latest and shortest of the multidimensional versions of the Symptom-Checklist 90-R.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Moriana E, Study Director — Universidad de Cordoba
Locations (1):
- Universidad de Córdoba, Córdoba, Córdoba, Spain

REFERENCES:
- [Derived] Galvez-Lara M, Corpas J, Vencesla JF, Moriana JA. Evidence-Based Brief Psychological Treatment for Emotional Disorders in Primary and Specialized Care: Study Protocol of a Randomized Controlled Trial. Front Psychol. 2019 Jan 8;9:2674. doi: 10.3389/fpsyg.2018.02674. eCollection 2018. PMID 30671005